CLINICAL TRIAL: NCT06068348
Title: Collection of Human Blood for Development of Liquid Biopsy Assay
Brief Title: Liquid Biopsy Collection Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00003221
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Chaperonin-Containing TCP-1; Circulating Tumor Cells; CCT; CTC
Keywords: Healthy
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to develop a liquid biopsy approach for detection of circulating tumor cells (CTC) that could be used in place of the more invasive and potentially risky methods of tissue biopsy. The aims of the project are: (a) determine whether the Chaperonin-Containing TCP-1 (CCT) chaperonin can used to identify rare cancer cells in blood, and (b) establish whether the cancer cells detected using the CCT chaperonin for identification have invasive or metastatic potential.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age greater than or equal to 18 and less than or equal to 80 years.

Exclusion Criteria:

* Adults unable to give informed consent
* Individuals who are not yet adults (infants, children, teenagers; under the age of 18)
* Individuals who weigh less than 110 lbs (as standard clinically advised to not give blood)
* Pregnant women (due to hormonal changes in blood)
* Prisoners
* Persons reporting a current microbial (bacterial, viral, or fungal) infections
* Persons reporting that they are current taking antibiotic medications
* Persons with body temperatures above 99oF (indicating a fever)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The researchers anticipate that the sample size of 60 will be adequate for statistical analysis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To determine if the biomarker, Chaperonin-Containing TCP-1 (CCT), can be used to detect circulating tumor cells (CTC) in blood. | 3 years

SECONDARY OUTCOMES:
To determine if the CCT chaperonin can provide information on the metastatic potential of CTC. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Annette Khaled, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States